CLINICAL TRIAL: NCT04654702
Title: A Multi-center, Prospective, Observational Study to Evaluate Therapeutic Effectiveness and Safety of Monterizine Cap in Patients With Asthma and Perennial Allergic Rhinitis.
Brief Title: Observational Study to Evaluate Therapeutic Effectiveness and Safety of Monterizine Cap.
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-MONT-OS-01
Record Dates: First submitted 2020-11-17; First posted 2020-12-04 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Perennial Allergic Rhinitis; Asthma
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigator examines the past prescription patterns and the reasons for the change of prescription to Monterizine capsules for Perennial Allergic Rhinitis patients with Asthma who will be taking Monterizine capsules to treat allergic rhinitis.

After being given Monterizine capsules, Investigator evaluates the therapeutic effectiveness and safety for 3 months (or 6 months).

DETAILED DESCRIPTION:
A Multi-center, Prospective, Observational Study

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 15 years
2. Perennial allergic rhinitis patients with asthma who will be prescribed Monterizine capsules to treat allergic rhinitis
3. Patients who provided a signed written informed consent form

Exclusion Criteria:

1. Highly sensitive patients to ingredients of Monterizine capsules, hydroxyzine or piperazine derivatives
2. Patients with renal failure(CLCR,10ml/min) and hemodialysis patients
3. A female who is pregnant, may be pregnant, or is lactating
4. Patients with genetic problems like Galactose intolerance, Lapp lactase deficiency or Glucose-galactose malabsorption

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 3,000 patients
Sampling Method: Probability Sample
Enrollment: 2671 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
The change in the average of TNSS at the point of Period 1 (recommended 3 Month(-1 Month)) as compared to baseline | 3 Month
  The change in the average of TNSS at the point of Period 1 (recommended 3 Month(-1 Month)) as compared to baseline.
  *TNSS: Total symptom scores for nasal congestion, sneezing, runny nose and nasal itching during the daytime in the past week

SECONDARY OUTCOMES:
The change in the average of TNSS at the point of Period 2(recommended 6Month(±1Month)) as compared to baseline | 6Month
  The change in the average of TNSS at the point of Period 2(recommended 6Month(±1Month)) as compared to baseline
The change in the therapeutic satisfaction at the point of Period 1 (recommended 3Month(-1Month)), Period 2(recommended 6Month(±1Month)) as compared to baseline | 3Month,6Month
  The change in the therapeutic satisfaction at the point of Period 1 (recommended 3Month(-1Month)), Period 2(recommended 6Month(1±Month)) as compared to baseline.
  *Therapeutic satisfaction : overall satisfaction with the treatment of allergic rhinitis for the past month. A possible scale is then: "Very Satisfied", "Satisfied", "Neutral", "Dissafistied", "Very Dissatisfied"
The change in the quality of life at the point of Period 1 (recommended 3Month(-1Month)), Period 2(recommended 6Month(±1Month)) as compared to baseline | 3Month,6Month
  The change in the quality of life at the point of Period 1 (recommended 3Month(-1Month)), Period 2(recommended 6Month(±1Month)) as compared to baseline.
  *Evaluate the quality of life with KARQLQ (Korean allergic rhinitis-specific quality of life questionnaire: 10 questions in regular activities at home and work, daily life disturbance and other symptoms)in the past week.
The change in the medication compliance at the point of Period 1 (recommended 3Month(-1Month)), Period 2(recommended 6Month(±1Month)) as compared to baseline | 3Month,6Month
  The change in the medication compliance at the point of Period 1 (recommended 3Month(-1Month)), Period 2(recommended 6Month(±1Month)) as compared to baseline.
  *Assessing the medication compliance for the last 30 days; compliance⪴80%, non-compliance<20%
Occurrence and frequency of adverse events | 6Month
  Occurrence and frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Byoung-Whui Choi, Principal Investigator — 59 institutions including Chung-Ang University Hospital
Locations (1):
- 59 institutions including Chung-Ang University Hospital, Seoul, South Korea